CLINICAL TRIAL: NCT03094546
Title: Effect of Polyamine-enriched Dietary Supplementation on Cognitive Function and Biomarkers in Elderly Individuals With Subjective Cognitive Decline
Brief Title: Polyamine-enriched Diet in Elderly Individuals With Subjective Cognitive Decline
Acronym: SmartAge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Freie Universität, Institute of Biology/Genetic, Berlin, Germany (Unknown); Karl-Franzens-Universität, Institute of Molecular Biosciences, Graz, Austria (Unknown)
Responsible Party: Principal Investigator, Claudia Schwarz, Postdoctoral Researcher, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SmartAge
Record Dates: First submitted 2017-03-14; First posted 2017-03-29 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Subjective Cognitive Decline (SCD)
Keywords: subjective cognitive decline; Alzheimer's disease, dementia; dietary supplement; polyamine; prevention; treatment; lifestyle; memory; autophagy
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Polyamines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyamine supplementation (Experimental): Intervention: Dietary Supplement (Polyamine supplementation): 750 mg wheat germ extract
  Interventions: Dietary Supplement: Polyamine
- Placebo (Placebo Comparator): Intervention: Dietary Supplement Placebo: 750 mg cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Polyamine — 12 months of polyamine supplementation (6 capsules/day)
  Arms: Polyamine supplementation
Dietary Supplement: Placebo — 12 months of placebo intake (6 capsules/day)
  Arms: Placebo

SUMMARY:
The overall objective of this study is to examine the effect of polyamine supplementation on cognitive performance and further characterization of individuals with subjective cognitive decline.

DETAILED DESCRIPTION:
Memory abilities are known to decline during aging, a process that is accelerated in pathological conditions like mild cognitive impairment (MCI) and Alzheimer's disease (AD), all of which are a growing public-health concern with devastating social and economical effects. Polyamines supplementation and corresponding up-regulation of autophagy (i.e., cellular protein degradation pathways) may be a key target of intervention against age-related memory decline. The study will investigate whether a polyamine-enriched dietary supplementation (through capsule intake) could provide positive effects on cognitive function and biomarkers of elderly individuals (60-90 years old) with subjective cognitive decline (SCD).

ELIGIBILITY:
Inclusion Criteria:

* Cognitive healthy individuals with subjective memory decline and self-reported concerns
* 60-90 years old
* No manifest dementia (DSM-IV criteria)
* No limitations in activities of daily living
* Capacity for consent

Exclusion Criteria:

* Gluten, histamine or wheat seedling intolerance
* Severe neurological, internal or psychological diseases
* Advanced heart or respiratory diseases, severe arteriosclerosis, untreated thyroid disease or diabetes
* Malignant tumors, current or past history
* Brain tumors, stroke
* Disorders that impair attention
* Dementia
* Coagulation disorder, Marcumar
* Drug abuse or alcohol dependency
* Current polyamine substitution

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change in Memory performance from neuropsychological test | change from baseline after 12 month (Prior to intervention (baseline T0) and after 12 months)
  Comparing memory function in subjects with polyamine intake and placebo treatment assessed prior to intervention (pre) vs. 12 month post intervention

SECONDARY OUTCOMES:
Change in Cognitive Function (from extended neuropsychological test battery) | change from baseline after 12 month
  Comparing cognitive function in subjects with polyamine intake and placebo treatment assessed prior to intervention (pre) vs. 12 month post intervention
Change in polyamine concentration | change from baseline after 12 month
  comparing polyamine concentration derived from blood plasma assessed prior to intervention (pre) vs. 12 month post intervention
Change in inflammation | change from baseline after 12 month
  comparing inflammation markers derived from blood plasma assessed prior to intervention (pre) vs. 12 month post intervention
Change in Brain imaging biomarkers | change from baseline after 12 month
  Multimodal analysis of biomarkers, regarding structural, functional, and perfusion-related plasticity, derived from magnet resonance imaging
Change in Autophagy processes | change from baseline after 12 month
  Evaluate autophagy processes through muscle biopsy assessed prior to intervention (pre) vs. 12 month post intervention
Change in Autophagy processes | change from baseline after 12 month
  Evaluate autophagy processes through blood parameters assessed prior to intervention (pre) vs. 12 month post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floeel, Prof, Principal Investigator — Charité - Universitätsmedizin Berlin, Greifswald Universitätsmedizin; Dietmar Schmitz, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité University Medicine Berlin, CCM, Department of Neurology,, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eisenberg T, Knauer H, Schauer A, Buttner S, Ruckenstuhl C, Carmona-Gutierrez D, Ring J, Schroeder S, Magnes C, Antonacci L, Fussi H, Deszcz L, Hartl R, Schraml E, Criollo A, Megalou E, Weiskopf D, Laun P, Heeren G, Breitenbach M, Grubeck-Loebenstein B, Herker E, Fahrenkrog B, Frohlich KU, Sinner F, Tavernarakis N, Minois N, Kroemer G, Madeo F. Induction of autophagy by spermidine promotes longevity. Nat Cell Biol. 2009 Nov;11(11):1305-14. doi: 10.1038/ncb1975. Epub 2009 Oct 4. PMID 19801973
- [Background] Gupta VK, Scheunemann L, Eisenberg T, Mertel S, Bhukel A, Koemans TS, Kramer JM, Liu KS, Schroeder S, Stunnenberg HG, Sinner F, Magnes C, Pieber TR, Dipt S, Fiala A, Schenck A, Schwaerzel M, Madeo F, Sigrist SJ. Restoring polyamines protects from age-induced memory impairment in an autophagy-dependent manner. Nat Neurosci. 2013 Oct;16(10):1453-60. doi: 10.1038/nn.3512. Epub 2013 Sep 1. PMID 23995066
- [Background] Ibe S, Kumada K, Yoshida K, Otobe K. Natto (fermented soybean) extract extends the adult lifespan of Caenorhabditis elegans. Biosci Biotechnol Biochem. 2013;77(2):392-4. doi: 10.1271/bbb.120726. Epub 2013 Feb 7. PMID 23391920
- [Background] Minois N, Carmona-Gutierrez D, Madeo F. Polyamines in aging and disease. Aging (Albany NY). 2011 Aug;3(8):716-32. doi: 10.18632/aging.100361. PMID 21869457
- [Background] Schaeffer V, Lavenir I, Ozcelik S, Tolnay M, Winkler DT, Goedert M. Stimulation of autophagy reduces neurodegeneration in a mouse model of human tauopathy. Brain. 2012 Jul;135(Pt 7):2169-77. doi: 10.1093/brain/aws143. Epub 2012 Jun 10. PMID 22689910
- [Background] Soda K, Dobashi Y, Kano Y, Tsujinaka S, Konishi F. Polyamine-rich food decreases age-associated pathology and mortality in aged mice. Exp Gerontol. 2009 Nov;44(11):727-32. doi: 10.1016/j.exger.2009.08.013. Epub 2009 Sep 6. PMID 19735716
- [Background] Soda K, Kano Y, Sakuragi M, Takao K, Lefor A, Konishi F. Long-term oral polyamine intake increases blood polyamine concentrations. J Nutr Sci Vitaminol (Tokyo). 2009 Aug;55(4):361-6. doi: 10.3177/jnsv.55.361. PMID 19763038
- [Background] Tiboldi A, Lentini A, Provenzano B, Tabolacci C, Hoger H, Beninati S, Lubec G. Hippocampal polyamine levels and transglutaminase activity are paralleling spatial memory retrieval in the C57BL/6J mouse. Hippocampus. 2012 May;22(5):1068-74. doi: 10.1002/hipo.22016. Epub 2012 Mar 30. PMID 22467251
- [Derived] Schwarz C, Benson GS, Horn N, Wurdack K, Grittner U, Schilling R, Marschenz S, Kobe T, Hofer SJ, Magnes C, Stekovic S, Eisenberg T, Sigrist SJ, Schmitz D, Wirth M, Madeo F, Floel A. Effects of Spermidine Supplementation on Cognition and Biomarkers in Older Adults With Subjective Cognitive Decline: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2213875. doi: 10.1001/jamanetworkopen.2022.13875. PMID 35616942
- [Derived] Wirth M, Schwarz C, Benson G, Horn N, Buchert R, Lange C, Kobe T, Hetzer S, Maglione M, Michael E, Marschenz S, Mai K, Kopp U, Schmitz D, Grittner U, Sigrist SJ, Stekovic S, Madeo F, Floel A. Effects of spermidine supplementation on cognition and biomarkers in older adults with subjective cognitive decline (SmartAge)-study protocol for a randomized controlled trial. Alzheimers Res Ther. 2019 May 1;11(1):36. doi: 10.1186/s13195-019-0484-1. PMID 31039826